CLINICAL TRIAL: NCT00389896
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Balanced, Three-Way Crossover Study to Evaluate the Efficacy of Simvastatin Therapy in Elevating HDL-C Levels in Patients With Type 2 Diabetic Dyslipidemia and Low HDL-C
Brief Title: A Crossover Study to Evaluate the Efficacy of Simvastatin in Elevating HDL-C Levels in Patients With Type 2 Diabetes (0733-216)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0733-216; 2006_536
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: HDL Cholesterol
MeSH Terms: interventions — Duration of Therapy

INTERVENTIONS:
Drug: MK0733 / Duration of Treatment: 18 Weeks
Drug: Comparator: placebo (unspecified) / Duration of Treatment: 18 Weeks

SUMMARY:
The purpose of this study is to see how well simvastatin raises HDL levels in patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has stable Type 2 diabetes mellitus at Visit 1.
* Patient meets screening criteria based on Visit 1 lab tests

Exclusion Criteria:

* Patient is pregnant, breastfeeding, or at risk of becoming pregnant
* Patient has heart disease, uncontrolled high blood pressure, or other significant disease
* Patient is taking prohibited medication(s) and is unable to stop taking them for the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-07-26 (Actual); Primary Completion 2002-10-04 (Actual); Study Completion 2002-10-04 (Actual)

PRIMARY OUTCOMES:
HDL-C raising effects after 6 weeks | 6 weeks

SECONDARY OUTCOMES:
Effect on other lipids and lipoproteins at 6 weeks | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Miller M, Dobs A, Yuan Z, Battisti WP, Palmisano J. The effect of simvastatin on triglyceride-rich lipoproteins in patients with type 2 diabetic dyslipidemia: a SILHOUETTE trial sub-study. Curr Med Res Opin. 2006 Feb;22(2):343-50. doi: 10.1185/030079906X80521. PMID 16466606
- [Background] Miller M, Dobs A, Yuan Z, Battisti WP, Borisute H, Palmisano J. Effectiveness of simvastatin therapy in raising HDL-C in patients with type 2 diabetes and low HDL-C. Curr Med Res Opin. 2004 Jul;20(7):1087-94. doi: 10.1185/030079904125004105. PMID 15265253